CLINICAL TRIAL: NCT00338195
Title: Assessment and Treatment of Caffeine Dependence
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Roland Griffiths, Professor, Department of Psychiatry, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPR01-05-04-03; R01DA001147 (NIH)
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2013-03-07 (Estimated); Status verified 2013-03

CONDITIONS: Self-identified Problematic Caffeine Use; DSM-IV Substance Dependence as Applied to Caffeine
Keywords: Caffeine dependence; Caffeine withdrawal

ARMS (1):
- Delayed intervention control (No Intervention)
  Interventions: Behavioral: Individualized caffeine cessation instructions

INTERVENTIONS:
Behavioral: Individualized caffeine cessation instructions — Intervention is described in the protocol

SUMMARY:
Recent research has established that some individuals report that they are unable to cease caffeine use, despite feeling that caffeine is posing a health risk or causing significant impairment in their daily activities. Despite the high rates of unsuccessful efforts to cease or control caffeine use in the population, there has been little research on the parameters of successful caffeine reduction and no research on caffeine cessation.

The goals of the study are as follows:

1. evaluate the applicability of DSM-IV dependence criteria for self-reported problematic caffeine use.
2. evaluate characteristics (e.g, co-morbid psychopathology) of individuals who report that they have had difficulty quitting caffeine use on their own and who are seeking treatment for caffeine use.
3. test the efficacy of a caffeine reduction treatment administered to individuals who would like to quit/reduce caffeine use, but have found it difficult to do so in the past.

DETAILED DESCRIPTION:
Recent research has established that some individuals report that they are unable to cease caffeine use, despite feeling that caffeine is posing a health risk or causing significant impairment in their daily activities. Despite the high rates of unsuccessful efforts to cease or control caffeine use in the population, there has been little research on the parameters of successful caffeine reduction and no research on caffeine cessation.

The goals of the study are as follows:

1. evaluate the applicability of DSM-IV dependence criteria for self-reported problematic caffeine use.
2. evaluate characteristics (e.g, co-morbid psychopathology) of individuals who report that they have had difficulty quitting caffeine use on their own and who are seeking treatment for caffeine use.
3. test the efficacy of a caffeine reduction treatment administered to individuals who would like to quit/reduce caffeine use, but have found it difficult to do so in the past.

Individuals will be recruited from the community via flyers, newspaper and radio advertisements. Those who are eligible will be invited to come to the Behavioral Pharmacology Research Unit. After consent is obtained (consent form A), a series of questionnaires will be completed (e.g., demographics, caffeine history, medical and psychiatric history, mood) followed by a structured clinical interview which will assess for a caffeine dependence syndrome and other psychopathology, as defined by the DSM-IV.

Afterwards, individuals who meet criteria will be offered the opportunity to receive assistance to reduce or quit using caffeine. Those who consent (Consent form B) to enroll in the second phase of the project will be randomly assigned to one of two conditions: 1. immediate treatment 2. wait-list control treatment. The conditions will be identical with the exception of the 6 week delay for one group. The treatment will consist of a brief individual counseling session, individualized caffeine tapering instructions, and a take home booklet. Participants return to BPRU at 6 weeks, 12 weeks, and 26 weeks post treatment to complete follow-up assessments. Participants will be assessed via telephone at 2 weeks and 52 weeks post-treatment. Follow- up measures will consist of self-reported caffeine use, biological measures of caffeine exposure (saliva), mood, and withdrawal questionnaires, and circumstances surrounding lapse incidences.

Inclusion criteria:

1. Consume >100mg caffeine per day
2. 18-65 years old
3. Medically healthy
4. Self-reported problem with caffeine use.

Exclusion criteria:

1. Pregnancy
2. Current dependence on alcohol or illicit drugs.

Risks and Benefits: The study procedures do not involve significant risk aside from the minor risk associated with a possible loss of confidentiality. Overall, this study will provide information about the occurrence of caffeine dependence syndrome as defined by the DSM-IV and the consumer demand for behavioral treatments for caffeine dependence. Furthermore, we will test a brief intervention for caffeine dependence. Presently there are no standard or empirically validated treatments for problematic caffeine use. Participants may benefit by receiving free assistance to reduce or cease their caffeine use. Society will benefit to the extent that successfully treating problematic caffeine use allows individuals to function more effectively.

Safety Monitoring: The principal investigator will review data any reports of untoward effects or possible adverse events.

ELIGIBILITY:
Inclusion Criteria:

1. Consume >100mg caffeine per day
2. 18-65 years old
3. Medically healthy
4. Self-reported problem with caffeine use.

Exclusion Criteria:

1. Pregnancy
2. Current dependence on alcohol or illicit drugs.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2001-05; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
self-reported caffeine use | as described in protocol

SECONDARY OUTCOMES:
biological measures of caffeine use | as described in protocol
mood questionnaires | as described in protocol

CONTACTS AND LOCATIONS:
Overall Officials: Roland R Griffiths, Ph.D., Principal Investigator — Professor, Johns Hopkins University School of Medicine
Locations (1):
- Behavioral Biology Research Center, Johns Hopkins Bayview, Baltimore, Maryland, United States